CLINICAL TRIAL: NCT00510536
Title: A Phase 4 Study to Assess the Practical Management of Mild to Moderate Arthritic or Arthralgic Events in Patients With Chronic Plaque Psoriasis Receiving Efalizumab
Brief Title: Treatment of Mild to Moderate Joint Pain in Patients With Chronic Plaque Psoriasis Receiving Efalizumab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Probity Medical Research (Network)
Responsible Party: Probity Medical Research, Probity Medical Research
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P07-104
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Last update posted 2009-04-10 (Estimated); Status verified 2009-04

CONDITIONS: Arthritis; Arthralgia
Keywords: Psoriasis, arthritis, arthralgia
MeSH Terms: conditions — Arthritis; Arthralgia; Psoriasis | interventions — Acetaminophen; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Acetaminophen — dose to be determined by investigator
Drug: NSAID — dose to be determined by investigator

SUMMARY:
The purpose of this study is to evaluate tolerability and effectiveness of conventional treatment for mild to moderate arthritic or arthralgic symptoms while subjects are being treated with efalizumab for psoriasis.

DETAILED DESCRIPTION:
The study objective is to demonstrate that mild to moderate arthritis or arthralgia may be controlled using conventional therapy while being treated with efalizumab, without loss of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Females cannot become pregnant while participating in study.
* Have a history of plaque psoriasis for at least 6 months.
* Receiving or about to receive efalizumab for the treatment of chronic plaque psoriasis.
* Have mild to moderate arthritis or arthralgia occurring while on treatment with efalizumab or untreated mild to moderate arthritis or arthralgia present at the time of initiating treatment with efalizumab.

Exclusion Criteria:

* Previous systemic treatment with biologics other than efalizumab, within 3 months.
* Treatment with any systemic corticosteroids or intra-articular corticosteroid injection, cyclosporine or methotrexate within 28 days.
* Any previous treatment with chlorambucil or cyclophosphamide.
* Have active tuberculosis or are currently receiving treatment or prophylactic therapy for tuberculosis.
* Have other serious disorders; such as, congestive heart failure, prior or current history of blood dyscrasia, or central nervous system demyelinating disorders.
* Has a sensitivity, intolerance, or history of gastrointestinal bleeding associated with diclofenac, indomethacin, and/or ibuprofen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

SECONDARY OUTCOMES:
The proportion of subjects who sustain or improve their psoriasis in response to efalizumab. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kim Papp, MD, PhD, Principal Investigator — K. Papp Clinical Research Inc.
Locations (1):
- K. Papp Clinical Research Inc., Waterloo, Ontario, Canada